CLINICAL TRIAL: NCT04125784
Title: Lipid Profile and Diabetes Risk of HIV Patients Treated by Austrian HIV -Physicians: a 7 Year Follow up Study
Brief Title: Lipid Profile and Diabetes Mellitus in People With HIV
Status: Completed | Type: Observational
Sponsor: Moritz Oberndorfer (Other)
Collaborators: Merck Gesellschaft mbH, Austria (Industry)
Responsible Party: Sponsor-Investigator, Moritz Oberndorfer, Researcher, Medical University of Vienna
Organization: Medical University of Vienna (Other)
Other Study IDs: V2_02082019
Record Dates: First submitted 2019-10-09; First posted 2019-10-14 (Actual); Last update posted 2023-03-31 (Actual); Status verified 2023-03

CONDITIONS: HIV Infections; Dyslipidemias; Diabetes Mellitus; Cardiovascular Risk Factor
Keywords: HIV; HIV infection; Dyslipidaemia; Diabetes mellitus; Diabetes mellitus type 2; Cardiovascular Risk factor; Lipid profile; Austria; HIV related treatment; Antiretroviral therapy; Follow-up Study
MeSH Terms: conditions — HIV Infections; Dyslipidemias; Diabetes Mellitus; Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Lipid-profile: The cohort includes male and female patients diagnosed and confirmed HIV diagnosis who receive HIV related treatment in an extramural setting. All patients are adults (older than 18 years old) and have participated in the original study in 2014.

SUMMARY:
Traditional risk factors for cardiovascular diseases have been shown to have an even higher impact in the HIV infected population. The original study from 2014 was a cross sectional study into the prevalence of cardiovascular risk factors (namely, dyslipidaemia and diabetes mellitus) in people living with HIV (PLWHIV) in Austria. The aim of this follow up study is to see the progression of our study sample and to see what prevalence levels may be found after 7 years. This epidemiological evaluation is conceptualized to document real life major cardiovascular risk factors of HIV-infected patients, focusing on lipid profiles and diabetes mellitus risk and to compare with the baseline values from the original study.

DETAILED DESCRIPTION:
Background: In developed countries, an increase in cardiovascular events and related mortality has been seen; even more prominent in people living with HIV (PLWHIV) as compared to non-HIV control groups. Studies have shown dyslipidaemia and diabetes mellitus type 2 as important risk factors for cardiovascular diseases in PLWHIV.

The original study by this group in 2014 was a cross sectional study into the prevalence of cardiovascular risk factors (dyslipidaemia and diabetes mellitus) in PLWHIV in Austria and identified characteristics associated with these two risk factors. In that previous study dyslipidaemia was diagnosed in 46.3% of cases and half of all the study participants showed an increased insulin resistance. Eight persons (1.6%) fulfilled the criteria for diabetes mellitus type 2.

Purpose: The aim of this follow up study is to see the progression of our study sample and to see what prevalence levels may be found after 7 years. Additionally, a look into previously identified characteristics associated with dyslipidaemia and diabetes mellitus type may provide valuable insight into the temporal effects. Finally, examining resource use this population in terms of medications can provide insights into current practice and its associated costs in Austria, as well as an estimate of the added medication cost of dyslipidaemia and diabetes mellitus type 2 in this population.

It is our aim to close the existing knowledge gap on the role of dyslipidaemia and diabetes mellitus on cardiovascular risk among PLWHIV in Austria. Therefore, the investigation will be carried out by using routine data within minimum additional effort to the study team. The data obtained may serve as a base for future decisions on treatment of the Austrian HIV population.

Study details: Our epidemiologic evaluation documents real life major cardiovascular risk factors of HIV-infected patients, focusing on lipid profiles and diabetes mellitus risk. The gathered data from approximately 450 originally enrolled patients will be compared with the baseline values analysed in the original study in 2014.

Data collection: Dataset definitions and the minimum dataset will be determined by the study authors. Parameters used and documented must match those that were taken in the original study. These were specified in the case report form (CRF). The data collection and preparation will be done by a student of the Medical University of Vienna (Department of Social and Preventive Medicine) as a part of the graduate thesis.

Enrolment Strategy: Patients will be recruited through the original study sites (2 extramural HIV clinics in Vienna). Original patient lists will be screened through the official Mortality Register of the Statistics Austria, where patients who have died during the follow up period will be identified. Additionally, other patients who decline participation will be asked to give reasons of declining participation.

Data Validation and Data quality: Accurate data are crucial contributors to informative statistical analyses. Missing data will not be systematized.

Quality Control: Source documentation and data accuracy will be verified by site visit(s) in 1 randomly selected site after termination of the enrolment period. 10% of case report forms of the reviewed site will be randomly selected for monitoring.

ELIGIBILITY:
Inclusion Criteria:

* Only Participants who participated in the previous study
* Adult (older than 18 years)
* male and female patients diagnosed and confirmed HIV diagnosis, given written informed consent

Exclusion Criteria:

* No participation in the original study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population includes only participants who participated in the original study from 2014. These patients are all patients who receive HIV related treatment in an extramural setting and visited their ÖGNÄ-HIV physician for routine control in Vienna/Austria. The original inclusion criteria were: adult (older than 18 years) male and female patients diagnosed and confirmed HIV diagnosis, given written informed consent.
Sampling Method: Non-Probability Sample
Enrollment: 450 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2023-02-28 (Actual)

PRIMARY OUTCOMES:
Changes in dyslipidemia prevalence from baseline - total cholesterol | 7 years
  Total cholesterol values will be analyzed by an authorized laboratory
Changes in dyslipidemia prevalence from baseline- triglycerides | 7 years
  Triglyceride values will be analyzed by an authorized laboratory
Changes in dyslipidemia prevalence from baseline - HDL-cholesterol | 7 years
  HDL-Cholesterol values will be analyzed by an authorized laboratory
Changes in dyslipidemia prevalence from baseline - Apolipoprotein B | 7 years
  Apolipoprotein B values will be analyzed by an authorized laboratory
Changes in dyslipidemia prevalence from baseline - LDL-cholesterol | 7 years
  a. LDL will be calculated using the Friedewald formula. As the Friedewald formula does not work in case of triglycerides > 300, in these patients only non-HDL-C will be used.
Changes in dyslipidemia prevalence from baseline - Non-HDL-Cholesterol | 7 years
  Non-HDL-Cholesterol will be calculated additionally.
Changes from baseline in diabetes mellitus type II prevalence | 7 years
  The diabetes mellitus prevalence will be assessed through patient history (checking for a diabetes mellitus type II diagnosis since baseline)

SECONDARY OUTCOMES:
Description of risk profile for cardiovascular events in the sample population | at follow up recruitment, Day 0
  The cardiovascular risk will be assessed through the European Society of Cardiology (ESC) calculator. Therefore, the risk profile for cardiovascular events will be assessed through documentation of risk factors (sex, age, smoking status, history of diabetes, hypertension, dyslipidaemia, previous cardiovascular events, other comorbidities) and laboratory parameters on the CRF by the investigator.
Changes from baseline in drug utilization for PLWHIV | 7 years
  Drug utilization will be assessed through documentation on the CRF by the investigator
Prevalence of diabetes mellitus type 2 in correlation to the prescribed antiretroviral regime during the follow up time | 7 years
  Diabetes mellitus type 2 will be assessed from patient history
Changes from baseline in the lipid profile of patients in correlation to prescribed antiretroviral regime | 7 years
  Lipid profile will be assessed with laboratory parameters (total cholesterol, triglycerides, HDL, Apolipoprotein B). LDL will be calculated using the Friedewald formula, additionally, non-HDL-Cholesterol (Non-HDL-C) will be calculated . As the Friedewald formula does not work in case of triglycerides > 300, in these patients only Non-HDL-C will be used.
Changes from baseline in therapy prescriptions of patients who were found to have hyperlipidaemia during first study in 2014 | 7 years
  Therapy prescriptions will be assessed through documentation of the patient's medication on the CRF by the investigator.
Documentation of any major cardiovascular events (stroke or heart attack) | during 7 years
  Cardiovascular events (stroke or heart attack) will be assessed through documentation on the CRF by the investigator.
Incidence of diabetes mellitus type 2 in patients who were diagnosed found to be insulin resistant in the first study in 2014 | 7 years
  Self reported diagnosis or presence of diabetes type 2 medication as noted in the CRF
Changes from baseline in therapeutic regimes within those patients who were identified as having diabetes mellitus type 2 in the first study in 2014 | 7 years
  Therapeutic regimes will be assessed through documentation of the patient's medication on the CRF by the investigator.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas E Dorner, MD, MPH, Principal Investigator — Medical University of Vienna
Locations (1):
- Schalk:Pichler Gruppenpraxis, Vienna, Austria

IPD SHARING:
Plan to Share IPD: Undecided
Anonymised and limited data set may be given to other researchers upon request from the principal investigator, following compliance of the Data Security Department of the Medical University of Vienna.